CLINICAL TRIAL: NCT06732206
Title: The Effect of Solution-Focused Approach on the Self-Control and Substance Use Risk Level of Nursing Students with Substance Use Risk
Brief Title: Substance Use Risk and Solution-Focused Approach
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ufuk DOĞAN (Other)
Responsible Party: Sponsor-Investigator, Ufuk DOĞAN, Lecturer PhD, Hasan Kalyoncu University
Organization: Hasan Kalyoncu University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2023/69
Record Dates: First submitted 2024-06-29; First posted 2024-12-13 (Actual); Last update posted 2024-12-13 (Actual); Status verified 2024-12

CONDITIONS: Self Efficacy
Keywords: Substance Use; Solution Focused Approach; Addiction; Tendency
MeSH Terms: conditions — Substance-Related Disorders; Behavior, Addictive

STUDY DESIGN:
Intervention Model Description: pretest - posttest experimental study with control group
Masking Description: It will be reported that the reasons for being included in the group are taken by a random method.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental Group (Experimental): The "short solution-oriented program" intervention group will be applied for 6 weeks, a total of 7 lesson hours.
  Interventions: Other: Short Solution Focused Approach Program
- Control Group (No Intervention)

INTERVENTIONS:
Other: Short Solution Focused Approach Program — It will be a psychoeducational approach aimed at developing preventive and protective properties against addiction.
  Arms: Experimental Group

SUMMARY:
Although substance abuse is the subject of serious struggles on the basis of individuals and countries, its rate of spread cannot be stopped and it creates an agenda with new people added every day. Substance addiction, which not only creates physiological problems in individuals, but also affects human health in every aspect with psychological and social problems, adversely affects the health status of individuals as well as their families and environments. The best way to get rid of addiction is to never start. Therefore, our study focused on preventing addiction, not addiction. After applying the Substance Use Tendency Scale and Self-Control Scale to university students, an intervention and control group will be formed. Solution Focused Approach program will be applied to the intervention group. At the end of the program, post-tests will be applied to the intervention and control groups.

DETAILED DESCRIPTION:
First of all, the Substance Use Tendency Scale (MDAS) and personal information form will be applied to the nursing students of the Faculty of Health Sciences, which consists of 750 people. A high score in any of the BCAS subscales indicates a tendency towards addiction. After this, students with a tendency will be determined. After the power analysis is performed, the appropriate number of samples will be determined. Finally, participants will be assigned to the intervention/control group by randomization. A substance use prevention psychoeducation program based on a solution-focused approach will be applied to the experimental group in 7 sessions for 6 weeks. No intervention will be made to the control group. At the end of psychoeducation, posttests will be collected from the experimental and control groups.

ELIGIBILITY:
The criteria for inclusion in the research at the stage;

* Being an active student registered as a nursing student at Fırat University
* Volunteering to participate in the research.
* Not receiving any psychological counseling and treatment
* Getting a sufficiently high score in any of the sub-dimensions according to the Substance Use Risk Profile Scale
* Not being diagnosed with substance abuse or substance abuse Exclusion criteria from the study at Phase I;
* Not complying with the principle of volunteering
* Getting a low score in all sub-dimensions according to the Substance Use Risk Profile Scale
* Being diagnosed with substance abuse or substance abuse

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 40 (Actual)
Dates: Start 2023-07-01 (Actual); Primary Completion 2023-11-01 (Actual); Study Completion 2024-06-30 (Actual)

PRIMARY OUTCOMES:
Changes in Students' Substance Use Risk Levels | 3 month period
  The scale developed by Woicik et al. (2009) and showing good psychometric properties in non-clinical samples was validated and reliability-tested in Turkish by Uygun et al. (2019). It is a 23-item (4-point Likert scale: 1 strongly disagree, 4 strongly agree) measurement tool. The scale has four subdimensions: hopelessness/self-discontent, impulsivity, sensation seeking, and anxiety sensitivity. The Cronbach's alpha value is determined to be 0.728. If at least one of the subscale scores is found to be high, it indicates a high risk of substance use in the individua
"Changes in the Self-Control Levels of Students at Risk of Substance Use | 3 month period
  The Self-Control Scale (SCS): The scale was developed by Rosenbaum in 1980. It measures how well individuals can use their existing control behaviors to solve problems they encounter in daily life. The Turkish validity and reliability studies were conducted by Duyan, Gülden, and Gelbal in 2012. The scale aims to estimate individuals' mental skills in controlling psychological and physiological responses such as anxiety, anger, and pain; delaying short-term satisfaction; initiating problem-solving processes; and self-efficacy perception. The scale consists of 3 sub-dimensions: Restorative Self-Control, Experiential Self-Control, and Renewing Self-Control, with a total of 36 items. Participants are asked to select one of the options prepared in a 6-point Likert type ranging from "Completely fits me +3" to "Completely does not fit me -3" in response to the questions. Higher scores on the scale indicate higher levels of self-control. The Cronbach's Alpha value was found to be 0.809.

CONTACTS AND LOCATIONS:
Overall Officials: Ufuk Doğan, PhD, Principal Investigator — Hasan Kalyoncu University
Locations (1):
- Ufuk Doğan, Elâzığ, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No